CLINICAL TRIAL: NCT05049642
Title: Effect of Chitosan-N-acetylcysteine (Lacrimera®) on Subjective Pain Sensation in Corneal Abrasion: a Pilot Study
Brief Title: Effect of Chitosan-N-acetylcysteine on Subjective Pain Sensation in Corneal Abrasion
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Medical device expired
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Principal Investigator, Vienna Institute for Research in Ocular Surgery
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Lacrimera Erosio
Record Dates: First submitted 2021-09-01; First posted 2021-09-20 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Eye Diseases
MeSH Terms: conditions — Eye Diseases

STUDY DESIGN:
Intervention Model Description: Patients will either be randomized to group 1 (instillation of 1 drop of C-NAC) or group 2 (no instillation of C-NAC) in a 1:1 fashion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Patients will either be randomized to group 1 (instillation of 1 drop of C-NAC) or group 2 (no instillation of C-NAC) in a 1:1 fashion. Afterwards one drop of C-NAC will be instilled into the study eye of group 1. 1 hour after treatment VAS and the symptom questionnaire will be performed repeatedly in both groups. Both groups will receive antibiotic ointment bandages and antibiotic eye drops for 5 days. Patients assigned to group 1 will receive Lacrimera® for home treatment over the following 5 days. 1 drop of Lacrimera® is supposed to be installed into the eye 20 minutes prior to installation of the respective antibiotic eye drops or ointments.
  Interventions: Device: Lacrimera
- Group 2 (No Intervention): Both groups will receive antibiotic ointment bandages and antibiotic eye drops for 5 days.

INTERVENTIONS:
Device: Lacrimera — A new preservative-free formulation of eye drops consists of a novel biopolymer, chitosan-N-acetylcysteine (C-NAC; Lacrimera®, Croma-Pharma GmbH, Leobendorf, Austria), which electrostatically binds to the mucine layer of the tear film forming a glycocalyx-like structure.
  Arms: Group 1

SUMMARY:
Aim of this study is to investigate the effect of Chitosan-N-acetylcysteine (C-NAC; Lacrimera®, Croma-Pharma GmbH, Leobendorf, Austria) in patients with corneal abrasion less than one third of the corneal surface on subjective pain sensation.

DETAILED DESCRIPTION:
Commonly, standard of care for corneal abrasion is topical antibiotics. Bandage contact lenses may be used in addition, which significantly decrease pain sensation in a vast majority of patients. Recently, a new preservative-free agent consisting of a novel biopolymer, Chitosan-N-acetylcysteine (C-NAC; Lacrimera®, Croma-Pharma GmbH, Leobendorf, Austria) has been approved for the treatment of dry eye syndrome (DES). This agent electrostatically binds to the mucine layer of the tear film, forming a glycocalyx-like structure. In an animal model, the beneficial effect of Chitosan-N-Acetylcysteine on recovery time has been observed. Aim of this study is to investigate the effect of Chitosan-N-acetylcysteine (C-NAC; Lacrimera®, Croma-Pharma GmbH, Leobendorf, Austria) in patients with corneal abrasion less than one third of the corneal surface on subjective pain sensation. It will further explore the extend of corneal healing after use of Lacrimera® over 5 days in those patients initially treated with Lacrimera®.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 years
* Corneal abrasion less than one third of the cornea

Exclusion Criteria:

* Ocular surgery within prior 3 months in the affected eye
* Ocular injury within prior 3 months before abrasion in the affected eye
* Ocular herpes of eye or eyelid within prior 3 months
* Active ocular infection
* Active ocular inflammation or history of chronic, recurrent ocular inflammation within prior 3 months
* Ocular surface abnormality that may compromise corneal integrity
* Presence of diseases that reduce experience of pain (e.g. Diabetes mellitus)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
VAS difference | 1 hour
  VAS difference between before application and one hour after instillation between the two groups

SECONDARY OUTCOMES:
Relative defect size difference | 7 days +/- 2 days
  Relative defect size difference as measured by fluorescein slit lamp photography between the visits between the two groups
Relative defect depth difference | 7 days +/- 2 days
  Relative defect depth difference as measured by AS-OCT at 1-week visit compared to baseline between the two groups
Size of haze | 7 days +/- 2 days
  Size of haze at 1 week visit between the two groups
VAS difference | 7 days +/- 2 days
  VAS difference at the one-week visit between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, PrimUnivPrDr, Principal Investigator — Vienna Institute for Research in Ocular Surgery
Locations (1):
- Vienna Institute for Research in Ocular Surgery, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No